CLINICAL TRIAL: NCT01249742
Title: Sugarsquare. Focus on the Adolescent: Digital Treatment of Type 1 Diabetes Through the Internet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Dr. C. Verhaak, Radboud University Nijmegen, Medical Center
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007.13.003
Record Dates: First submitted 2010-11-22; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; adolescent; online intervention; psychosocial; quality of life
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Internet intervention — Our intervention, Sugarsquare, is a secured treatment environment only accessible by patients of the KDCN and members of the treatment team. Sugarsquare consists of two main sections. The first section is a semi-public setting on which adolescents can exchange experiences with their diabetes (care) through a forum and a real time chat-application. All patients and treatment team members can see all messages posted here. The second section consists of patients' individual pages with treatment overview and an application for private interaction with the treatment team. Patients can only access their own individual page; treatment team members can access pages of all patients. Sugarsquare is a secured webpage, accessible only through computers equipped with the right certificate (access device) and by using the appointed username-password combination.

SUMMARY:
Background

The treatment of diabetes is multidisciplinary. Alignment of care of the various professional disciplines is, however, not always optimal. This can lead to confusion about treatment interventions and behavioral advices. In adolescence, good fine-tuned care is of extreme importance because of the difficulties in regulation of the disease in this phase of life (Snoek, 2004). These difficulties are due to biological changes but also to socio-psychological developmental changes. The adolescents' psychological development demands more autonomy and responsibility for the diabetes (care) by the adolescent. The social development can conflict with the treatment regime, because of the adolescents' social needs (ADA, 2001; Houdijk, 1998; Snoek, 2004). In this study the investigators assess whether an interactive website, on which adolescents with diabetes and their treatment team can communicate, leads to better alignment of care and better control over the disease.

Intervention

The diabetes has great impact on the adolescents' everyday life. Finding a balance between more autonomy, participating in social life with (healthy) peers and control of the disease is difficult and seems to act as a thread during this phase in life.

This can lead to questions and uncertainty at any given moment. The interactive website provides the adolescent access to information and to his or her individual treatment plan and advices fitted to his or her condition and life. The adolescent can pose questions at any given moment through the online forum and their personal treatment page. Since the treatment team answers the question within a day, fit between diabetes care and adolescents' everyday life is optimized.

Research question

Does an online interactive treatment environment, on which adolescents with diabetes can communicate with their treatment team, lead to better fit of care and to better disease control?

ELIGIBILITY:
Inclusion Criteria:

* adolescents aged 12 and older;
* diagnosed with diabetes mellitus;
* receiving regular outpatient hospital-delivered diabetes care provided by the Children's Diabetes Center Nijmegen (CDCN)

Exclusion Criteria:

* adolescents who were unable to read questionnaires because of language, or cognitive problems were excluded

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Patients' Evaluation of Quality of Care | T0: baseline (1 month prior to acces to intervention); T1: (6 months following T0); T2: (12 months following T0).
  Participants' appreciation of our diabetes care was assessed using the Patients' Evaluation of Quality of Diabetes care (PEQ-D; Pouwer & Snoek, 2002). This questionnaire consists of 14 items, such as: 'The amount of information I receive from the doctor is…'. The adolescent is asked to answer by means of a 5-point lykert scale varying from 1) bad to 5) excellent.

SECONDARY OUTCOMES:
Health Related Quality of Life | T0: baseline (1 month prior to acces to intervention); T1: (6 months following T0); T2: (12 months following T0).
  Health-related quality of life was measured by means of the PedsQl 3.0 diabetes module (Varni, 2004). The Dutch translation was used, which shows good psychometric properties for clinical application in pediatric diabetes care (de Wit, 2008). The questionnaire consists of 28 items and can be subdivided into five subscales; diabetes symptoms, treatment barriers, treatment adherence, worry, and communication. Example of item: 'I feel hungry' (subscale diabetes symptoms). Al items can be answered using a 5-point lykert scale, varying from 0 (never) to 4 (almost always).
Adolescents' disease knowledge | T0: baseline (1 month prior to acces to intervention); T1: (6 months following T0); T2: (12 months following T0).
  Diabetes knowledge was measured using the Diabetes Knowledge Questionnaire (Fitzgerald, 1998). This questionnaire has shown to have good psychometric properties (Fitzgerald, 1998). The questionnaire was translated in Dutch especially for this study. The final Dutch version, DKT-NL, consisted of 21 multiple choice questions, such as 'sings of ketoacidosis include… '. Possible answers were: a) shakiness, b) sweating, c) vomiting (right answer), d) low blood glucose .
Confidence In Diabetes Selfcare | T0: baseline (1 month prior to acces to intervention); T1: (6 months following T0); T2: (12 months following T0).
  Participants' self-efficacy was determined through use of the Confidence In Diabetes Selfcare questionnaire (CIDS; van de ven, 2004). The questionnaire contains 20 items, all referring to the perceived ability to perform diabetes self-care tasks. All items are preceded by "I believe I can… ," and can be answered on a 5-point lykert scale, varying from 1) "No, I am sure I cannot" to 5) "Yes, I am sure I can"). An example is "I believe I can… adjust my insulin when I am sick".
Glycemic control (HbA1c) | T0: baseline (1 month prior to acces to intervention); T1: (6 months following T0); T2: (12 months following T0).
  Patients' Glycemic control was derived from their files. 'Old' HbA1c values were converted to new HbA1c values using the calculator of the Dutch Diabetes Federation (NDF, 2010). New HbA1c values were used in the analyses.
Degree of use of intervention | T1 (6 months following start of intervention)
  The degree of use of our intervention was measured by frequency of use of adolescents of different applications. We therefore logged all action of adolescents on Sugarsquare. Examples of variables are number of page views, number of posted messages on the forum, number of attended chat sessions and number of started discussions with professional caregivers. Table 3 gives insight in all actions included in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Emiel Boogerd, MSc., Principal Investigator — Radboud University Nijmegen, Medical Center; Chris Verhaak, Dr., Principal Investigator — Radboud University Nijmegen, Medical Center; Kees Noordam, Dr., Principal Investigator — Radboud University Nijmegen, Medical Center
Locations (1):
- Children's Diabetes Center Nijmegen, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Boogerd EA, Noordam C, Kremer JA, Prins JB, Verhaak CM. Teaming up: feasibility of an online treatment environment for adolescents with type 1 diabetes. Pediatr Diabetes. 2014 Aug;15(5):394-402. doi: 10.1111/pedi.12103. Epub 2013 Dec 18. PMID 24350732